CLINICAL TRIAL: NCT01516216
Title: Randomized, Double-Blind, Phase II Trial of Vitamin D Supplementation in Patients With Previously Untreated Metastatic Colorectal Cancer
Brief Title: Study of Vitamin D in Untreated Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Kimmie Ng, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-436
Record Dates: First submitted 2012-01-13; First posted 2012-01-24 (Estimated); Results first posted 2022-03-23 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: previously untreated
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol; Bevacizumab; Fluorouracil; Leucovorin; Oxaliplatin; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy + Standard Dose Vitamin D (Active Comparator): FOLFOX-bevacizumab: intravenously on Day 1 (+/- 7 days) of every two-week cycle per institutional standards + 400 IU vitamin D3 orally once daily
  Participants were treated until disease progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: FOLFOX + bevacizumab; Dietary Supplement: Vitamin D
- Chemotherapy + Higher Dose (Active Comparator): FOLFOX-bevacizumab: intravenously on Day 1 (+/- 7 days) of every two-week cycle per institutional standards + 8000 IU daily x 2 weeks as loading dose, followed by 4000 IU daily as maintenance dose.
  Participants were treated until disease progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: FOLFOX + bevacizumab; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: FOLFOX + bevacizumab
  Other Names: 5-FU (5-fluorouracil); Leucovorin; Oxaliplatin (Eloxatin); Bevacizumab (Avastin)
Dietary Supplement: Vitamin D

SUMMARY:
This is a prospective, randomized, double-blind phase II trial to evaluate the efficacy and safety of two doses of vitamin D supplementation in combination with standard chemotherapy in participants with previously-untreated metastatic colorectal adenocarcinoma.

DETAILED DESCRIPTION:
In this research study, the investigators are comparing standard and higher dose Vitamin D treatment when given in combination with standard treatment for metastatic colorectal cancer. Standard treatment includes the chemotherapy combination of 5-FU, Leucovorin and Oxaliplatin (FOLFOX) with bevacizumab.

Participants will be randomized into one of the study groups-Arm A: Vitamin D (standard dose of 400 IU/day), FOLFOX and Bevacizumab or Arm B: Vitamin D (higher dose of 8000 IU/day for 2 weeks followed by 4000 IU/day), FOLFOX and Bevacizumab.

Study Treatment (A cycle of treatment is 14 days):

Vitamin D

Cycle 1: You will take two capsules of Vitamin D orally, once a day (at the same time), every day. Participants randomized to Arm A will be taking one capsule with 400 IU of Vitamin D and one capsule with placebo (pills with no medicine) so that neither you nor your doctor will know what group you have been assigned to. Participants randomized to Arm B will be taking two capsules of 4000 IU each.

Subsequent Cycles: You will take one capsule orally, once a day (at the same time), every day. Participants randomized to Arm A will be taking one capsule with 400 IU of Vitamin D. Participants randomized to Arm B will be taking one capsule with 4000 IU of Vitamin D.

FOLFOX and bevacizumab

FOLFOX and bevacizumab will be given intravenously (IV, through a vein in your arm) on Day 1 of every cycle for all participants in both Arms A and B. The infusions will take several hours, in addition to your doctor's visit, so you should plan on being in clinic most of the day. Note that the 5-FU is given bolus on day 1 (given as one dose), and is then given as a continuous IV infusion over 2 days. You will need to have a port-a-cath placed. A port-a-cath is a medical device that is placed under the skin. The continuous infusion is delivered by a pump that is inserted into the port-a-cath. The pump will be carried in a pouch that you can hook around your waist. Arrangements will be made for you to have the pump disconnected after 2 days. You may need to return to clinic to have it disconnected.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the colon or rectum that is metastatic or locally advanced (unresectable)
* Measurable disease
* KRAS wild-type and KRAS mutant patients are eligible
* No prior systemic treatment for advanced or metastatic colorectal cancer is allowed
* No prior radiotherapy to more than 25% of bone marrow
* No surgery or major biopsy within 4 weeks of randomization
* Paraffin-embedded and/or snap-frozen tumor tissue samples must be available

Exclusion Criteria:

* Not pregnant or breastfeeding
* No prior chemotherapy, systemic therapy or investigational agent
* No concurrent use of other anti-cancer therapy
* No known brain metastases
* No history of other malignancies except adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, curatively treated lobular or ductal carcinoma in situ of the breast or other cancer curatively treated with no evidence of disease for more than 3 years prior to randomization
* No regular use of vitamin D supplements greater than 2000 IU per day in the past year
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to 5-FU, capecitabine, oxaliplatin, leucovorin, bevacizumab and/or vitamin D3
* No significant history of bleeding events, pre-existing bleeding diathesis, coagulopathy or gastrointestinal perforation
* No arterial thrombotic events within 6 months of randomization
* No serious non-healing wound, ulcer or bone fracture
* No history of uncontrolled hypertension
* No clinically significant peripheral neuropathy
* No predisposing colonic or small bowel disorders in which the symptoms are uncontrolled
* No uncontrolled seizure disorder or active neurological disease
* No pre-existing hypercalcemia
* No known active hyperparathyroid disease
* No regular use of thiazide diuretics
* No malabsorption, uncontrolled vomiting or diarrhea
* No known co-morbid disease that would increase the risk of toxicity
* No use of chronic oral corticosteroid therapy or any other therapy that can cause vitamin D depletion
* No clinically significant cardiovascular disease
* No uncontrolled intercurrent illness
* No history of any medical or psychiatric condition or addictive disorder or laboratory abnormality that may increase the risks associated with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2012-04-13 (Actual); Primary Completion 2019-11-09 (Actual); Study Completion 2019-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimmie Ng, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (18):
- United States (18):
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Mountain States Tumor Institute- Fruitland, Fruitland, Idaho
  - Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Mountain States Tumor Institute- Nampa, Nampa, Idaho
  - Mountain States Tumor Institute- Twin Falls, Twin Falls, Idaho
  - The Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional Medical Center, Milford, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center in clinical affiliation with South Shore Hospital, South Weymouth, Massachusetts
  - New Hampshire Oncology Hematology-P.A., Concord, New Hampshire
  - New Hampshire Oncology Hematology-P.A., Hooksett, New Hampshire
  - New Hampshire Oncology Hematology-P.A., Laconia, New Hampshire
  - Dana-Farber/New Hampshire Oncology-Hematology, Londonderry, New Hampshire
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Background] Ng K, Nimeiri HS, McCleary NJ, Abrams TA, Yurgelun MB, Cleary JM, Rubinson DA, Schrag D, Miksad R, Bullock AJ, Allen J, Zuckerman D, Chan E, Chan JA, Wolpin BM, Constantine M, Weckstein DJ, Faggen MA, Thomas CA, Kournioti C, Yuan C, Ganser C, Wilkinson B, Mackintosh C, Zheng H, Hollis BW, Meyerhardt JA, Fuchs CS. Effect of High-Dose vs Standard-Dose Vitamin D3 Supplementation on Progression-Free Survival Among Patients With Advanced or Metastatic Colorectal Cancer: The SUNSHINE Randomized Clinical Trial. JAMA. 2019 Apr 9;321(14):1370-1379. doi: 10.1001/jama.2019.2402. PMID 30964527

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from April 2012 through November 2016.
Groups:
- Chemotherapy + Higher Dose Vitamin D: FOLFOX-bevacizumab: intravenously on Day 1 (+/- 7 days) of every two-week cycle per institutional standards + 8000 IU daily x 2 weeks as loading dose, followed by 4000 IU daily as maintenance dose.
  Participants were treated until disease progression, unacceptable toxicity or withdrawal for other reasons.
Period: Overall Study
Arm/Group | Chemotherapy + Standard Dose Vitamin D | Chemotherapy + Higher Dose Vitamin D
Started | 70 | 69
AE Evaluable (Participants who started treatment were evaluable for AEs however all participants were followed for death (all-cause mortality).) | 67 | 68
Response Evaluable (Participants who started treatment were evaluable for response if underwent >/=1 restaging scan.) | 62 | 66
Completed (Given treatment duration is not fixed, all participants are considered as 'Non Completed' and reason discontinued treatment provided.) | 0 | 0
Not Completed | 70 | 69
Not completed — Adverse Event | 2 | 4
Not completed — Disease Progression | 38 | 34
Not completed — Withdrawal by Subject | 9 | 11
Not completed — Potentially Curative Resection | 6 | 12
Not completed — Nonadherence | 2 | 3
Not completed — Physician Decision | 6 | 3
Not completed — Prolonged Treatment Delay | 5 | 1
Not completed — Intercurrent Illness | 1 | 0
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy + Standard Dose Vitamin D | Chemotherapy + Higher Dose Vitamin D | Total
Number analyzed (Participants) | 70 | 69 | 139
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 56 [50 to 64] | 54 [47 to 65] | 55 [24 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 28 | 60
  Male | 38 | 41 | 79
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 55 | 52 | 107
  Black | 6 | 4 | 10
  Asian | 1 | 0 | 1
  >1 race | 1 | 2 | 3
  Other | 7 | 11 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 70 | 69 | 139
ECOG performance status [Count of Participants; unit: Participants] — 0 - Fully active, able to carry on all pre-disease performance without restriction
  1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    0 | 40 | 29 | 69
    1 | 30 | 40 | 70
Primary Tumor Location [Count of Participants; unit: Participants]
  Right colon (cecum, ascending colon, hepatic flexure) | 19 | 16 | 35
  Transverse colon | 8 | 4 | 12
  Left colon (splenic flexure, descending colon, sigmoid, rectosigmoid, rectum) | 43 | 49 | 92
Primary tumor resected [Count of Participants; unit: Participants] | 21 | 26 | 47
Received prior adjuvant therapy [Count of Participants; unit: Participants] | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival (PFS)
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. Per RECIST 1.1 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
  Patients who discontinued treatment to pursue potentially curative resection were censored for progression-free survival at the time of surgery. Patients who had not experienced cancer progression or died were censored at their last known follow-up date.
Time Frame: Disease was evaluated every 4 cycles on treatment and off treatment every 8-16 weeks until PD or non-protocol therapy start if discontinued for reason other than PD. Participants were observed up to 28.5 months with maximum follow-up of 56.7 months.
Population: the analysis population is comprised of all randomized patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemotherapy + Standard Dose Vitamin D | Chemotherapy + Higher Dose Vitamin D
Number analyzed (Participants) | 70 | 69
Months | 11 [9.5 to 14] | 13 [10.1 to 14.7]
Statistical Analysis 1: Comparison: Chemotherapy + Standard Dose Vitamin D vs Chemotherapy + Higher Dose Vitamin D; Test type: Superiority; p = 0.07, Log Rank

2. Secondary Outcome: Median Overall Survival (OS)
Description: OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive. Patients who discontinued treatment to pursue potentially curative resection were censored for progression-free survival at the time of surgery. Patients who had not experienced cancer progression or died were censored at their last known follow-up date.
Time Frame: Participants were followed for survival by clinic visit or telephone every 3 months post-treatment discontinuation up to 36 months from the date that the last participant was enrolled. Median follow-up was 22.9 months with maximum 56.7 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Chemotherapy + Standard Dose Vitamin D | Chemotherapy + Higher Dose Vitamin D
Number analyzed (Participants) | 70 | 69
Months | 24.3 [20.3 to 32.4] | 24.3 [19.0 to 33.2]
Statistical Analysis 1: Comparison: Chemotherapy + Standard Dose Vitamin D vs Chemotherapy + Higher Dose Vitamin D; Test type: Superiority; p = 0.43, Log Rank

3. Secondary Outcome: Objective Response Rate
Description: The objective response rate (ORR) was defined as the percentage of participants achieving complete response (CR) or partial response (PR) based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease was evaluated every 4 cycles on treatment. Median (maximum) treatment duration was 7.3 (28.5) months.
Population: The analysis population is comprised of the response evaluable subset.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy + Standard Dose Vitamin D | Chemotherapy + Higher Dose Vitamin D
Number analyzed (Participants) | 62 | 66
percentage of participants | 63 [50 to 75] | 58 [45 to 70]
Statistical Analysis 1: Comparison: Chemotherapy + Standard Dose Vitamin D vs Chemotherapy + Higher Dose Vitamin D; Test type: Superiority; p = 0.27, Chi-squared

4. Secondary Outcome: Grade 3-5 Treatment-Related Neutropenia Toxicity Rate
Description: The percentage of treated participants experiencing grade 3-5 neutropenia with treatment attribution of possible, probable or definite based on Common Toxicity Criteria for Adverse Events version 4 (CTCAEv4) as reported on case report forms were counted.
Time Frame: AEs were evaluated at day 1 of each cycle on treatment and up to 30 days after the last dose. Maximum treatment duration is 28.5 months with median 7.3 months.
Population: The analysis population is comprised of the subset evaluable for adverse events.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy + Standard Dose Vitamin D | Chemotherapy + Higher Dose Vitamin D
Number analyzed (Participants) | 67 | 68
percentage of participants | 31 [21 to 44] | 35 [24 to 48]

5. Secondary Outcome: Number of Participants With Vitamin D Deficiency at Baseline
Description: Vitamin D deficiency was defined as plasma 25-hydroxyvitamin D [25(OH)D] level <20 ng/mL as measured in one batch per established methods by an independent laboratory.
Time Frame: Baseline
Population: The analysis population is comprised of the subset with evaluable plasma samples at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy + Standard Dose Vitamin D | Chemotherapy + Higher Dose Vitamin D
Number analyzed (Participants) | 61 | 63
Participants | 39 | 48
Statistical Analysis 1: Comparison: Chemotherapy + Standard Dose Vitamin D vs Chemotherapy + Higher Dose Vitamin D; Test type: Superiority; p = 0.68, Chi-squared

6. Secondary Outcome: Vitamin D Sufficiency Rate
Description: Percentage of participants that achieve Vitamin D sufficiency defined as plasma 25(OH)D >=30 ng/mL on treatment as measured in one batch per established methods by an independent laboratory.
Time Frame: Plasma samples were collected at 3 timepoints on treatment: first restaging (cycle 5, day 1), second restaging (cycle 9, day 1) and at treatment discontinuation. Median (maximum) treatment duration was 7.3 (28.5) months.
Population: The analysis population is comprised of the subset with evaluable plasma samples at each collection timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy + Standard Dose Vitamin D | Chemotherapy + Higher Dose Vitamin D
Number analyzed (Participants) | 61 | 63
percentage of participants | 9.8 [4.2 to 20.2] | 71.4 [59.2 to 81.2]

7. Secondary Outcome: Plasma 25-hydroxyvitamin D Levels
Description: Plasma 25-hydroxyvitamin D [25(OH)D] levels as measured in one batch per established methods by an independent laboratory.
Time Frame: Plasma samples were collected at 4 timepoints on study: baseline, first restaging (cycle 5, day 1), second restaging (cycle 9, day 1) and at treatment discontinuation. Median (maximum) treatment duration was 7.3 (28.5) months.
Population: The analysis population is comprised of the subset with evaluable plasma samples at each collection timepoint.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Chemotherapy + Standard Dose Vitamin D | Chemotherapy + Higher Dose Vitamin D
Number analyzed (Participants) | 61 | 63
ng/mL
  Baseline plasma 25(OH)D levels | 18.7 [13.5 to 22.7] | 16.1 [10.1 to 23.0]
  First restaging plasma 25(OH)D levels: number analyzed (Participants) | 50 | 54
  First restaging plasma 25(OH)D levels | 18.7 [16.1 to 22.5] | 32 [25.7 to 39.5]
  Second restaging plasma 25(OH)D levels: number analyzed (Participants) | 37 | 47
  Second restaging plasma 25(OH)D levels | 18.5 [16.0 to 22.6] | 35.2 [25.0 to 45.4]
  At treatment discontinuation plasma 25(OH)D levels: number analyzed (Participants) | 47 | 43
  At treatment discontinuation plasma 25(OH)D levels | 18.7 [13.9 to 23.0] | 34.9 [24.9 to 44.7]

8. Secondary Outcome: Hazard Ratio Between Baseline Plasma 25(OH)D Level and PFS
Description: Plasma 25-hydroxyvitamin D [25(OH)D] levels as measured in one batch per established methods by an independent laboratory. Plasma 25(OH)D Level is used as continuous data. PFS is estimated based on Kaplan-Meier method (see outcome measure 1). The PFS hazard ratio associated with one unit increase of 25()H)D.
Time Frame: Baseline Plasma 25(OH)D Level and up to 28.5m for evaluation of PFS.
Population: The analysis population is comprised of all participants with evaluable Plasma 25(OH)D Level samples at baseline.
Measure: Number (95% Confidence Interval); unit: hazard ratio
Groups:
- All Participants With Baseline Plasma 25 (OH) D Level: Evaluated prior to treatment.
Arm/Group | All Participants With Baseline Plasma 25 (OH) D Level
Number analyzed (Participants) | 124
hazard ratio | 1.00 [0.97 to 1.03]
Statistical Analysis 1: Comparison: All Participants With Baseline Plasma 25 (OH) D Level; Test type: Superiority; p = 0.9801, Chi-squared

9. Secondary Outcome: Hazard Ratio Between Baseline Plasma 25(OH)D Levels and OS
Description: Plasma 25-hydroxyvitamin D [25(OH)D] levels as measured in one batch per established methods by an independent laboratory. Plasma 25(OH)D Level is used as continuous data. OS is estimated based on Kaplan-Meier method (see outcome measure 2). The OS hazard ratio associated with one unit increase of 25()H)D.
Time Frame: Baseline Plasma 25(OH)D Level and up to maximum 56.7 months for evaluation of OS.
Population: The analysis population is comprised of all participants with evaluable Plasma 25(OH)D Level samples at baseline.
Measure: Number (95% Confidence Interval); unit: hazard ratio
Groups:
- All Participants of the Study: 70 were assigned FOLFOX-bevacizumab q 2 weeks + 400 IU vitamin D3 orally once daily, 69 were assigned FOLFOX-bevacizumab: intravenously on Day 1 (+/- 7 days) of every two-week cycle per institutional standards + 8000 IU daily x 2 weeks as loading dose, followed by 4000 IU daily as maintenance dose.
Arm/Group | All Participants of the Study
Number analyzed (Participants) | 124
hazard ratio | 0.995 [0.96 to 1.03]
Statistical Analysis 1: Comparison: All Participants of the Study; Test type: Superiority; p = 0.7444, Chi-squared

ADVERSE EVENTS:
Time Frame: AEs were evaluated at day 1 of each cycle on treatment and up to 30 days after the last dose. Maximum treatment duration is 28.5 months with median 7.3 months. All-Cause Mortality was assessed up to 56.7 months and Serious and Other (Not Including Serious) adverse events were assessed up to 29.5 months (the additional 30 days of monitoring included in the maximum treatment duration).
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Chemotherapy + Standard Dose Vitamin D | Chemotherapy + Higher Dose Vitamin D
All-Cause Mortality (participants affected / at risk) | 54/67 | 45/68
Serious Adverse Events (participants affected / at risk) | 39/67 | 47/68
Other Adverse Events (participants affected / at risk) | 65/67 | 67/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy + Standard Dose Vitamin D (N=67) | Chemotherapy + Higher Dose Vitamin D (N=68)
Anemia (Blood and lymphatic system disorders) | 4 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac disorders - Other (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 5 | 3
Non-cardiac chest pain (General disorders) | 1 | 0
General disorders and administration site conditions - Other (General disorders) | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 6 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Rectal perforation (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Lip infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2
Alkaline phosphatase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Cardiac troponin I increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 3
Neutrophil count decreased (Investigations) | 21 | 22
Platelet count decreased (Investigations) | 0 | 1
Weight loss (Investigations) | 0 | 2
White blood cell decreased (Investigations) | 4 | 4
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 6
Seizure (Nervous system disorders) | 1 | 0
Stroke (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal calculi (Renal and urinary disorders) | 1 | 0
Hypertension (Vascular disorders) | 10 | 9
Thromboembolic event (Vascular disorders) | 1 | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy + Standard Dose Vitamin D (N=67) | Chemotherapy + Higher Dose Vitamin D (N=68)
Ear pain (Ear and labyrinth disorders) | 0 | 1
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 36 | 34
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 4
Leukocytosis (Blood and lymphatic system disorders) | 6 | 4
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 3 | 8
Chest pain - cardiac (Cardiac disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 3 | 0
Pericardial effusion (Cardiac disorders) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 2 | 1
Sinus tachycardia (Cardiac disorders) | 7 | 11
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Cardiac disorders - Other (Cardiac disorders) | 1 | 1
Chills (General disorders) | 5 | 6
Edema face (General disorders) | 0 | 1
Edema limbs (General disorders) | 11 | 4
Facial pain (General disorders) | 0 | 2
Fatigue (General disorders) | 60 | 59
Fever (General disorders) | 12 | 10
Flu like symptoms (General disorders) | 1 | 2
Gait disturbance (General disorders) | 5 | 2
Infusion related reaction (General disorders) | 2 | 3
Irritability (General disorders) | 2 | 1
Localized edema (General disorders) | 1 | 0
Neck edema (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 11 | 9
Pain (General disorders) | 24 | 17
General disorders and administration site conditions - Other, specify (General disorders) | 12 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 9
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 6
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 1
Erythroderma (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 2
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 | 2
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 16 | 10
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 4
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 10 | 5
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 9 | 10
Abdominal distension (Gastrointestinal disorders) | 6 | 4
Abdominal pain (Gastrointestinal disorders) | 26 | 35
Anal hemorrhage (Gastrointestinal disorders) | 3 | 4
Anal pain (Gastrointestinal disorders) | 1 | 2
Ascites (Gastrointestinal disorders) | 1 | 1
Bloating (Gastrointestinal disorders) | 5 | 7
Cheilitis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 1
Colonic fistula (Gastrointestinal disorders) | 1 | 1
Colonic obstruction (Gastrointestinal disorders) | 1 | 1
Colonic perforation (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 33 | 42
Diarrhea (Gastrointestinal disorders) | 32 | 44
Dry mouth (Gastrointestinal disorders) | 5 | 0
Duodenal hemorrhage (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 7 | 16
Dysphagia (Gastrointestinal disorders) | 6 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0
Fecal incontinence (Gastrointestinal disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 9 | 4
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 | 5
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 5 | 3
Lip pain (Gastrointestinal disorders) | 3 | 0
Mucositis oral (Gastrointestinal disorders) | 30 | 19
Nausea (Gastrointestinal disorders) | 44 | 53
Oral dysesthesia (Gastrointestinal disorders) | 2 | 3
Oral hemorrhage (Gastrointestinal disorders) | 2 | 1
Oral pain (Gastrointestinal disorders) | 9 | 6
Rectal hemorrhage (Gastrointestinal disorders) | 5 | 7
Rectal pain (Gastrointestinal disorders) | 6 | 5
Rectal perforation (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Stomach pain (Gastrointestinal disorders) | 1 | 2
Tooth development disorder (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 19 | 28
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 21 | 18
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 3 | 3
Catheter related infection (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Lip infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 1
Nail infection (Infections and infestations) | 0 | 1
Papulopustular rash (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Rhinitis infective (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 3 | 0
Skin infection (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 2
Upper respiratory infection (Infections and infestations) | 4 | 5
Upper respiratory infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 4
Vulval infection (Infections and infestations) | 1 | 0
Infections and infestations - Other (Infections and infestations) | 1 | 7
Bruising (Injury, poisoning and procedural complications) | 3 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 7
Prolapse of intestinal stoma (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 2
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 3 | 1
Alanine aminotransferase increased (Investigations) | 16 | 12
Alkaline phosphatase increased (Investigations) | 22 | 24
Aspartate aminotransferase increased (Investigations) | 26 | 26
Blood bilirubin increased (Investigations) | 6 | 11
Carbon monoxide diffusing capacity decreased (Investigations) | 1 | 0
Cholesterol high (Investigations) | 2 | 0
Creatinine increased (Investigations) | 4 | 4
GGT increased (Investigations) | 0 | 1
Haptoglobin decreased (Investigations) | 0 | 1
Hemoglobin increased (Investigations) | 1 | 0
INR increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 9 | 4
Neutrophil count decreased (Investigations) | 18 | 19
Platelet count decreased (Investigations) | 34 | 29
Urine output decreased (Investigations) | 1 | 0
Weight gain (Investigations) | 1 | 2
Weight loss (Investigations) | 15 | 13
White blood cell decreased (Investigations) | 21 | 19
Investigations - Other (Investigations) | 16 | 21
Acidosis (Metabolism and nutrition disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 33 | 29
Dehydration (Metabolism and nutrition disorders) | 4 | 6
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 27 | 31
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 3
Hypernatremia (Metabolism and nutrition disorders) | 2 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 12 | 14
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 7
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 5
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 4 | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 8 | 18
Hyponatremia (Metabolism and nutrition disorders) | 10 | 11
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 5
ME133 (Metabolism and nutrition disorders) | 7 | 2
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 16
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 | 6
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 4 | 6
Cognitive disturbance (Nervous system disorders) | 1 | 0
Concentration impairment (Nervous system disorders) | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 12 | 9
Dysesthesia (Nervous system disorders) | 21 | 21
Dysgeusia (Nervous system disorders) | 17 | 12
Facial muscle weakness (Nervous system disorders) | 1 | 0
Glossopharyngeal nerve disorder (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 16 | 19
Lethargy (Nervous system disorders) | 0 | 1
Movements involuntary (Nervous system disorders) | 1 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 5 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 49 | 55
Presyncope (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 0 | 1
Sinus pain (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 2 | 5
Syncope (Nervous system disorders) | 1 | 1
Transient ischemic attacks (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 1
Vasovagal reaction (Nervous system disorders) | 0 | 1
Nervous system disorders - Other (Nervous system disorders) | 15 | 17
Blurred vision (Eye disorders) | 3 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 4 | 1
Scleral disorder (Eye disorders) | 0 | 1
Watering eyes (Eye disorders) | 2 | 2
Eye disorders - Other (Eye disorders) | 2 | 2
Agitation (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 12 | 13
Confusion (Psychiatric disorders) | 2 | 1
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 6 | 8
Insomnia (Psychiatric disorders) | 11 | 21
Personality change (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 2
Suicidal ideation (Psychiatric disorders) | 0 | 3
Psychiatric disorders - Other (Psychiatric disorders) | 1 | 4
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 14
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 | 24
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Hematuria (Renal and urinary disorders) | 7 | 4
Proteinuria (Renal and urinary disorders) | 6 | 12
Renal calculi (Renal and urinary disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 2
Urine discoloration (Renal and urinary disorders) | 1 | 2
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 7
Irregular menstruation (Reproductive system and breast disorders) | 1 | 0
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 3 | 1
Penile pain (Reproductive system and breast disorders) | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 2 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 1
Menopause (Reproductive system and breast disorders) | 1 | 0
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 2 | 0
Flushing (Vascular disorders) | 1 | 2
Hot flashes (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 27 | 30
Hypotension (Vascular disorders) | 3 | 7
Thromboembolic event (Vascular disorders) | 3 | 1
Thromboembolic event (Vascular disorders) | 3 | 3
Vascular disorders - Other (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/16/NCT01516216/Prot_SAP_000.pdf